CLINICAL TRIAL: NCT05043792
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study of TT-00920 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Dose of TT-00920 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TT00920US03
Record Dates: First submitted 2021-09-01; First posted 2021-09-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 (Low dose) (Active Comparator): TT-00920, orally, three times daily (t.i.d.) from Day 1 to Day 13 and once on Day 14.
  Interventions: Drug: TT-00920
- Dose 2 (High dose) (Active Comparator): TT-00920, orally, three times daily (t.i.d.) from Day 1 to Day 13 and once on Day 14.
  Interventions: Drug: TT-00920
- Placebo (Placebo Comparator): TT-00920 Placebo, orally, three times daily (t.i.d.) from Day 1 to Day 13 and once on Day 14.
  Interventions: Drug: TT-00920 Placebo

INTERVENTIONS:
Drug: TT-00920 — TT-00920 Tablets
  Arms: Dose 1 (Low dose); Dose 2 (High dose)
Drug: TT-00920 Placebo — TT-00920 Placebo Tablets
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multiple ascending dose escalation study of TT-00920 in healthy subjects.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multiple ascending dose escalation study of TT-00920 in healthy subjects. Each dosing cohort will be comprised of 10 randomized subjects dosed three times daily for 13 days and one time for 1 day. The study will consist of a Screening Period, an In-house Period and a Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Age ≥ 18.0 years and ≤ 55.0 years, male or female
* BMI between 18.0 and 30.0 kg/m2, inclusive, and weighs at least 50.0 kg
* No clinically significant findings in medical examination

Exclusion Criteria:

* Known hypersensitivity or allergy to lactose
* Vaccination with any live vaccine, or vaccination employing an mRNA platform within 28 days and/or vaccination with any inactivated vaccine within 7 days of study drug administration
* Impaired cardiac function including clinically significant arrhythmias or clinically significant abnormality
* HbA1c > 5.7 % at Screening
* Subject with a history of severe visual diseases; or visual changes
* Subject is unable to complete this study for other reasons or the Investigator believes that he or she should be excluded

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs and clinically relevant changes in safety parameters,e.g. clinical laboratory tests, 12-lead ECG, ophthalmological examination [Safety and tolerability] | 14 days
  * TEAE: Treatment emergent adverse events
  * Safety parameters: physical examinations, vital signs, clinical laboratory tests , 12-lead ECG in triplicate, cardiac Holter monitoring, visual tests and ophthalmological examinations

SECONDARY OUTCOMES:
Area under the plasma drug concentration versus time curve at steady state (AUC0-t, ss and AUC0-τ, ss) | 14 days
Maximum observed plasma concentration at steady state (Cmax, ss) | 14 days
Time corresponding to occurrence of Cmax,ss at steady state (Tmax, ss) | 14 days
Minimum observed plasma concentration at steady state (Cmin, ss) | 14 days
Trough plasma concentration (Ctrough) | 14 days
Accumulation ratio (Rac) | 14 days
Average concentration (Cav) | 14 days
Volume of distribution at steady state (Vz/F, ss) | 14 days
Clearance at steady state (CL/F, ss) | 14 days
Half-life at steady state (T1/2, ss) | 14 days

OTHER OUTCOMES:
Metabolite characterization in plasma and estimation | 14 days
  observed drug-related material in plasma to determine the presence of any metabolite >10%
Change in Biomarkers From Baseline to Day 14: cGMP (Pmol/mL) | 14 days
  cGMP: cyclic guanosine monophosphate
Utilization of PGx results | 14 days
  A pharmacogenomic (PGx) panel will be performed to test for genetic variations in genes related to drug response

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No